CLINICAL TRIAL: NCT06826989
Title: A Phase 1 Study to Evaluate the Absorption, Metabolism, and Excretion of [14C]MK-8527 in Healthy Adult Participants
Brief Title: A Study of MK-8527 in Healthy Adult Participants (MK-8527-013)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8527-013; MK-8527-013 (Other: MSD)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]MK-8527 (Experimental): Participants will receive a single oral dose of [14C]MK-8527 on Day 1
  Interventions: Drug: [14C]MK-8527

INTERVENTIONS:
Drug: [14C]MK-8527 — Oral Dose

SUMMARY:
The goal of this study is to learn how [14C]MK-8527 moves through a healthy person's body over time. Researchers will study how [14C]MK-8527 is absorbed by the body, broken down by the body, and how it leaves the body.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health
* Has a body mass index (BMI) of 18 to 32 kg/m^2

Exclusion Criteria:

* Has a history of cancer
* Has positive tests for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Cumulative Percentage of Total Radioactivity Recovered (fe) from Urine and Feces | At designated timepoints (up to approximately 5 weeks post-dose)
  Urine and fecal samples will be collected to determine the cumulative percentage of radioactivity recovered from both urine and feces.
Fe from Urine | At designated timepoints (up to approximately 5 weeks post-dose)
  Urine samples will be collected to determine the percent of total radioactivity recovered from urine.
Fe from Feces | At designated timepoints (up to approximately 5 weeks post-dose)
  Fecal samples will be collected to determine the percent of total radioactivity recovered from feces.
Plasma MK-8527: Area Under the Concentration-Time Curve from Time 0 to 24 Hours Post-dose (AUC0-24) | At designated timepoints (up to 24 hours post-dose)
  Plasma samples will be collected to determine the AUC0-24 of MK-8527.
Plasma MK-8527: Maximum Observed Concentration (Cmax) | At designated timepoints (up to approximately 14 days post-dose)
  Plasma samples will be collected to determine the Cmax of MK-8527.
Plasma MK-8527: Concentration at 24 Hours Post-dose (C24) | At designated timepoints (up to 24 hours post-dose)
  Plasma samples will be collected to determine the C24 of MK-8527.
Plasma MK-8527: Time of the Maximum Observed Concentration (Tmax) | At designated timepoints (up to approximately 14 days post-dose)
  Plasma samples will be collected to determine the Tmax of MK-8527.
Plasma Total Radioactivity: AUC0-24 | At designated timepoints (up to 24 hours post-dose)
  Plasma samples will be collected to determine the AUC0-24 of total radioactivity.
Plasma Total Radioactivity: Cmax | At designated timepoints (up to approximately 5 weeks post-dose)
  Plasma samples will be collected to determine the Cmax of total radioactivity.
Plasma Total Radioactivity: C24 | At designated timepoints (up to 24 hours post-dose)
  Plasma samples will be collected to determine the C24 of total radioactivity.
Plasma Total Radioactivity: Tmax | At designated timepoints (up to approximately 5 weeks post-dose)
  Plasma samples will be collected to determine the Tmax of total radioactivity.
Whole Blood Total Radioactivity: AUC0-24 | At designated timepoints (up to 24 hours post-dose)
  Whole blood samples will be collected to determine the AUC0-24 of total radioactivity.
Whole Blood Total Radioactivity: Cmax | At designated timepoints (up to approximately 5 weeks post-dose)
  Whole blood samples will be collected to determine the Cmax of total radioactivity.
Whole Blood Total Radioactivity: C24 | At designated timepoints (up to 24 hours post-dose)
  Whole blood samples will be collected to determine the C24 of total radioactivity.
Whole blood Total Radioactivity: Tmax | At designated timepoints (up to approximately 5 weeks post-dose)
  Whole blood samples will be collected to determine the Tmax of total radioactivity.
Cumulative Amount of Radioactivity Recovered from Urine | At designated timepoints (up to approximately 5 weeks post-dose)
  Urine samples will be collected to determine the cumulative amount of radioactivity recovered from urine.
Percent of Total Radioactive Dose Recovered from Urine | At designated timepoints (up to approximately 5 weeks post-dose)
  Urine samples will be collected to determine the percent of the total radioactive dose recovered from urine.
Cumulative Amount of Radioactivity Recovered from Feces | At designated timepoints (up to approximately 5 weeks post-dose)
  Fecal samples will be collected to determine the cumulative amount of radioactivity recovered from feces.
Percent of Total Radioactive Dose Recovered from Feces | At designated timepoints (up to approximately 5 weeks post-dose)
  Fecal samples will be collected to determine the percent of the total radioactive dose recovered from feces.
Total Number of Metabolites in Plasma that Represent at least 10% of the Dose of Radioactivity | At designated timepoints (up to approximately 5 weeks post-dose)
  Plasma samples will be collected at pre-specified timepoints and used to determine the total number of metabolites that represent at least 10% of the dose of radioactivity. Metabolites will be determined using liquid scintillation and high-resolution mass spectrometry.
Total Number of Metabolites in Urine that Represent at least 10% of the Dose of Radioactivity | At designated timepoints (up to approximately 5 weeks post-dose)
  Urine samples will be collected at pre-specified timepoints and used to determine the total number of metabolites that represent at least 10% of the dose of radioactivity. Metabolites will be determined using liquid scintillation and high-resolution mass spectrometry.
Total Number of Metabolites in Feces that Represent at least 10% of the Dose of Radioactivity | At designated timepoints (up to approximately 5 weeks post-dose)
  Fecal samples will be collected at pre-specified timepoints and used to determine the total number of metabolites that represent at least 10% of the dose of radioactivity. Metabolites will be determined using liquid scintillation and high-resolution mass spectrometry.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue the Study Due to an AE | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Fortea CRU Madison ( 0001), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com